CLINICAL TRIAL: NCT06094647
Title: Altitudes for Caregivers: A Pilot Study
Brief Title: Altitudes for Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-1676
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: Care Burden; Care Giving Burden; Caregiver Burnout; Caregiver Stress; Caregiver Wellbeing; Support, Family
Keywords: Digital Intervention; Social Media; Virtual Therapeutic Content; Virtual Educational Content; Supporters; Caregiving
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Altitudes Condition (Experimental): Approximately 30 individuals whose loved ones are experiencing FEP and receiving services from two of the five FEP clinics (OASIS and SHORE) will be recruited to participate in a digital platform, Altitudes, for 6 months as part of an adjunct service to the clinic's services. Participants will have access to and encouraged to use the educational and therapeutic content as well as the moderated online community network during their time engaging with the platform. They will be asked to complete a battery of measures at baseline, 3-months, and 6 months.
  Interventions: Device: Altitudes USA
- Treatment as Usual (No Intervention): Approximately 30 individuals whose loved ones are experiencing FEP and receiving services from three of the five FEP clinics (Encompass, Eagle, and AEGIS) will be recruited to participate in treatment as usual offered by their respective clinic. Participants will then be asked to complete the same battery of measures as the experimental group at baseline, 3-months, and 6 months.

INTERVENTIONS:
Device: Altitudes USA — Experimental participants will be onboarded to the digital platform, including the different spaces and how to use the site. The site includes educational and therapeutic content that is tailored to each individual and their current needs and experiences, including psychoeducation, supporting their loved one, self-care, social support, and so on. Further, the platform includes a moderated social media function, where users and family peer workers can post text, images, videos, and comments to connect and share their experiences. The site is monitored by graduated students and trained clinicians.
  Arms: Altitudes Condition

SUMMARY:
The objective of this study is to assess the acceptability and feasibility of Altitudes, a novel digital behavioral health and psychoeducational intervention for caregivers and supporters of individuals experiencing first episode psychosis. The investigators will evaluate acceptability and feasibility with up to 30 caregivers and supporters over the course of 6 months. Acceptability and usability will be assessed with various acceptability measures with the Altitudes caregivers and supporters, caregivers and supporters' engagement with the digital platform, and qualitative interviews with the Altitudes caregivers and supporters. The investigators will additional evaluate the impact of the platform on caregiver and supporter's psychological status, wellbeing, and social support, as measured via self-report questionnaires.

DETAILED DESCRIPTION:
Purpose: The purpose of the present study is to investigate the acceptability and feasibility of implementing a moderated online social media platform with therapeutic content, Altitudes, as a part of an adjunct services offered at first-episode psychosis (FEP) clinics across North Carolina, also known as coordinated specialty care (CSC) programs. Additionally, to further assess the secondary aims of impact on experiences, wellbeing, and support from the platform, the investigators will recruit a control group of caregivers and supporters from clinics that do not have access to or are piloting the digital platform.

Participants: Thirty parent or caregiver and supporter participants from OASIS and SHORE CSC clinics will be recruited for the Altitudes condition and 30 caregiver or supporter participants from Eagle, Encompass, AEGIS, We2Care, OASIS, and SHORE clinics will be recruited for the control condition.

Procedures (methods): All participants will be recruited over a 20-week to 28-week period at from the North Carolina's first episode psychosis (FEP) clinics. The Altitudes condition participants will be recruited from OASIS and SHORE, while the control participants will be recruited from the Eagle, Encompass, AEGIS, and We2Care in addition to OASIS and SHORE. Altitude participants will engaged with the digital platform, known as Altitudes, for approximately 6 months. Site usage information as well as feedback about their experience will be collected from these participants through the Altitudes platform. Site usage information (e.g., number of posts/comments made on the site, the number and types of 'Journeys' or 'Tracks' (psychoeducation and therapeutic content) completed by participants, etc.) will be collected automatically through the Altitudes platform. Before being given access to Altitudes, a research coordinator, family peer support specialist, or moderator will provide instructions and guidance for using the site (i.e., Altitudes onboarding). Experiences, wellbeing, and support measures will be collected at baseline, mid-treatment (~3 months) and post-treatment (~6 months) for the Altitudes participants. Additional feedback in the form of a qualitative interview will be collected from the Altitudes participants at the end of six months intervention.

As Altitudes involves psychoeducational and therapeutic content, this platform is considered an adjunct to the clinical care provided to caregivers and supporters by FEP clinics. As such, Altitudes participants will not be compensated for their involvement in the platform. Site usage information will be collected automatically through the Altitudes site. However, Altitudes participants will be compensated for providing feedback about their experience with Altitudes as well as for completing other assessments.

Finally, Altitudes will be monitored at least once daily by trained family peer support specialists, master's level clinicians, and/or graduate students with relevant clinical/research experience with individuals experiencing psychosis and their caregivers and supporters. Drs. David Penn and Kelsey Ludwig, trained clinical psychologists, will lead weekly supervision calls to ensure appropriate care and support of Altitudes participants involved in this project, to discuss case conceptualization and suggestions for engaging individuals in the platform, as well as to monitor any potential safety concerns.

The control participants will not engage with the Altitudes platform. They will be recruited from the Eagle, Encompass, AEGIS, and We2Care clinics primarily with the option to recruit from OASIS and SHORE as well from the family therapy and/or multi-family groups. They will meet with research staff at three time points (baseline, 3 months, and 6 months) to complete a battery of measures that mirror the measures completed by the Altitudes participant group. Control participants will be compensated for meeting with research staff and completing the battery of measures.

ELIGIBILITY:
Inclusion Criteria:

* Parent, caregiver, or supporter of a young person who is currently receiving treatment from a CSC program for FEP, or who have recently graduated from a CSC program
* Parent, caregiver, or supporter must be at least 18 years of age
* Participants recruited from Outreach and Support Intervention Services (OASIS) & Supporting Hope, Opportunities, Recovery and Empowerment (SHORE; i.e., two CSC programs in NC), as this is a pilot study, or Eagle, Encompass, AEGIS, We2Care, SHORE, or OASIS clinics for participants part of the control group
* Parent, caregiver, or supporter must have access to internet through a mobile phone, tablet, or computer

Exclusion Criteria:

* Parent, caregiver, or supporter is currently engaged in legal action against the loved one receiving services from the CSC program
* Parent, caregiver, or supporter does not speak English
* Parent, caregiver, or supporter is under 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Diana Perkins, MD, MPH, Principal Investigator — Univeristy of North Carolina, School of Medicine; Kelsey Ludwig, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication and provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Requesting investigator has appropriate approval (see above) and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The research team attempted to recruit participants for a treatment as usual condition, but the coordinated specialty care (CSC) programs that were encouraged to refer caregivers indicated that family members of young people with first episode psychosis (FEP) were not interested in completing assessments without the option of joining the Altitudes program (treatment condition). Therefore, no participants were enrolled into the Treatment as Usual Arm.
Period: Overall Study
Arm/Group | Altitudes Condition | Treatment as Usual
Started | 24 | 0
Completed | 24 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled into the Treatment as Usual Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Altitudes Condition | Treatment as Usual | Total
Number analyzed (Participants) | 24 | 0 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.38 (8.28) |  | 57.38 (8.28)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender Female | 17 |  | 17
  Cisgender Male | 6 |  | 6
  Transgender Female | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  | 2
  Not Hispanic or Latino | 21 |  | 21
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 2 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 20 |  | 20
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 |  | 24

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Summaries of Participant Experience in Post-Treatment Feedback
Description: This qualitative data will be collected post-treatment from Altitudes participants. Individual interviews will discuss usage of the platform and any feedback participants may have. Feedback from participants will be summarized to include common themes regarding likes and dislikes of the platform, implementation within the clinical setting, and participant ideas for future directions.
Time Frame: Up to 6 months
Population: No participants were enrolled into the Treatment as Usual Arm. Two participants elected not to complete the post-treatment interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 22 | 0
Participants
  Altitudes described as a valuable resource | 17 |
  Clinical moderator was a useful source of support | 17 |
  Life circumstances impacted engagement | 14 |
  Reduced participation due to life demands or intentional avoidance (e.g., topic of psychosis) | 9 |
  Altitudes platform was a space for connection, learning, hope, and/or normalizing their experiences | 18 |
  Therapy materials were appropriated and added to their knowledge/understanding/skills | 15 |
  Altitudes was easy to access, navigate, and use | 19 |
  Caregivers mentioned wanting notifications or reminders | 10 |
  Caregivers interested opportunities to meet other parents/carers | 7 |
  Caregivers note interest in or benefits to tailored supports (like individual therapy) | 7 |

2. Primary Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions (WAI-I) - Total Score
Description: The Working Alliance Inventory for Guided Internet Interventions (WAI-I) is a 12-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always." Possible scores are averaged across items and range from 1 to 5. Higher scores indicate greater therapeutic alliance. Reported value is the average value at month 6 minus the average value at month 3.
Time Frame: Month 3, Month 6
Population: No participants were enrolled into the Treatment as Usual Arm. All data collected are reported. Four participants elected not to complete the post-treatment assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.27 (0.58) |

3. Primary Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions (WAI-I) - Task and Goals Subscale
Description: The Working Alliance Inventory for Guided Internet Interventions (WAI-I) task and goals subscale is an 8-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores are averaged across items and range from 1 to 5. Higher scores indicate greater agreement between the therapist and client on tasks and goals.
Time Frame: Month 3, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.23 (0.74) |

4. Primary Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions (WAI-I) - Bond Subscale
Description: The Working Alliance Inventory for Guided Internet Interventions (WAI-I) is a 4-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores are averaged across items and range from 1 to 5. Higher scores indicate stronger bond with the supporting therapist
Time Frame: Month 3, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.35 (0.77) |

5. Primary Outcome: Mean Engagement With the Altitudes Platform
Description: The Altitudes platform passively collects engagement data, including the number of therapeutic education modules started and completed as well as any posts, reactions, or comments made on the platform. The investigators will provide mean and standard deviation scores for each site usage category, for the Altitudes group only. The data was collected continuously from baseline up to month 6 as a count of occurences with the mean engagement with the Altitudes platform computed across this time frame.
Time Frame: Baseline, Up to Month 6
Population: No participants were enrolled into the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: number of occurrences
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
number of occurrences
  Posts on community page | 2.92 (4.13) |
  Comments on Other Users' Posts | 9.79 (18.49) |
  Reactions to Other Users' Posts | 21.13 (33.98) |
  Comments on the Talk-it-Out Page (e.g., problem-solving) | 1.88 (2.76) |
  Posts on the Talk-it-Out Page (e.g., problem-solving) | 0.29 (0.46) |
  Reactions on the Talk-it-Out Page (e.g., problem-solving) | 3.54 (6.39) |
  Number of Calls Attended with Clinical Moderator | 5.71 (3.10) |
  Number of Meet-ups attended | 3.00 (1.92) |
  Number of Journey Steps (therapy content) | 16.25 (15.58) |
  Number of Explore Steps (therapy content) | 18.68 (18.03) |

6. Primary Outcome: Mean Change in Altitudes Health Care Climate Questionnaire (A-HCCQ) - Total Score
Description: The Altitudes Health Care Climate Questionnaire is a 15-item scale. Answers are on a 7-point Likert scale (1-7) with options "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 15 to 105 with higher scores reflecting better perceptions of their relationship with Altitudes moderators.
Time Frame: Month 3, Month 6
Population: Only participants who have completed both assessments have been included in this analysis. No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 19 | 0
score on a scale | 0.12 (0.61) |

7. Primary Outcome: Mean Change in Altitudes Perceived Competence Scale (A-PCS) - Total Score
Description: The Altitudes Health Care Climate Questionnaire is a 4-item scale. Answers are on a 7-point Likert scale with options "Not at all true"[1], "Somewhat true"[4], "Very true"[7] with a sliding scale between answers. Possible scores range from 4 to 28. Higher scores indicate stronger perceived competence and ability in using the Altitudes platform.
Time Frame: Month 3, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.19 (0.99) |

8. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Overall Impressions of Platform Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The overall impressions of the platform scale is three 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 3 to 21. Higher scores indicate better overall impressions of the Altitudes platform.
Time Frame: Month 3, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.50 (1.25) |

9. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Perception of Other Platform Users Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The perception of other platform users subscale is four 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 4 to 28. Higher scores indicate better perception of interactions with other Altitudes participants.
Time Frame: Month 3, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.30 (1.16) |

10. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Safety and Confidentiality Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The safety and confidentiality subscale is two 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 2 to 14. Higher scores indicate higher perceived safety and confidentiality when using the platform.
Time Frame: Month 3, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.25 (1.03) |

11. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Moderation and Peer Support Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The moderation and peer support subscale is three 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 3 to 21. Higher scores indicate higher regard of the moderators and peer support on the Altitudes platform.
Time Frame: Month 3, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.18 (1.19) |

12. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Barriers to Use Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The barriers to use subscale is six 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 6 to 42. Lower scores indicate less issues with barriers to engaging with the platform.
Time Frame: Month 3, Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 20 | 0
score on a scale | 0.53 (0.32) |

13. Secondary Outcome: Mean Change in University of California, Los Angeles (UCLA) Loneliness Scale - Total Score
Description: The UCLA Loneliness scale is a 20-item scale. Answers are on a 4-point scale with options "I often feel this way," "I sometimes feel this way," "I rarely feel this way," and "I never feel this way." Possible scores range from 20 to 80. Higher scores reflect worse outcomes (greater feelings of loneliness). The UCLA Loneliness Scale is a part of the PhenX Toolkit.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.01 (0.11) |

14. Secondary Outcome: Mean Change in Multidimensional Scale of Perceived Social Support - Total Score [Alternative Form for Altitudes Participants, Original Form for Control Group]
Description: The Multidimensional Scale of Perceived Social Support Survey is a 16-item scale. Answers are on a 7-point scale with options ranging from "very strongly disagree" to "very strongly agree". Possible scores range from 16 to 112. Higher scores reflect higher feelings of social support (more perceived social support).
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.01 (0.11) |

15. Secondary Outcome: Mean Change in the Experience of Caregiving Inventory (ECI) - Total Score
Description: The ECI Scale is a 66-item scale. Answers are on a 5-point scale starting at 0 with options "never," "rarely," "sometimes," "often," and "nearly always". Possible scores range from 0 to 264 after appropriate items have been reversed scored. Higher scores indicate greater feelings of preparedness for caregiving whereas lower scores reflect feeling less prepared to provide caregiving.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 2.54 (3.1) |

16. Secondary Outcome: Mean Change in the Experience of Caregiving Inventory (ECI) - Positive Experience Subscales
Description: The ECI Scale is a 66-item scale. Answers are on a 5-point scale starting at 0 with options "never," "rarely," "sometimes," "often," and "nearly always". The positive experience subscale is 14 items with possible scores range from 0 to 56. Higher scores indicate greater feelings of preparedness and experiences with caregiving.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 3.73 (1.48) |

17. Secondary Outcome: Mean Change in the Experience of Caregiving Inventory (ECI) - Negative Experiences Subscale
Description: The ECI Scale is a 66-item scale. Answers are on a 5-point scale starting at 0 with options "never," "rarely," "sometimes," "often," and "nearly always". The negative experience subscale is 52 items with possible scores range from 0 to 208. Higher scores reflect feeling less prepared to provide caregiving and more negative experiences in caregiving.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 1.34 (4.72) |

18. Secondary Outcome: Mean Change in Family Questionnaire of Expressed Emotion - Total Score
Description: The Family Questionnaire (FQ) is a 20-item, self-administered questionnaire that measures expressed emotion status (criticism and emotional over involvement (EOI)) of family members toward patients with mental illness. The FQ has two subscales: critical comments, and EOI. Each item is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The FQ is scored by adding together the ratings from the individual items. Possible scores range from 20 to 80 with higher scores indicating greater levels of expressed emotion.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.05 (0.18) |

19. Secondary Outcome: Mean Change in Family Questionnaire of Expressed Emotion - Critical Comments Subscale
Description: The Family Questionnaire (FQ) is a 20-item, self-administered questionnaire that measures expressed emotion status (criticism and emotional over involvement (EOI)) of family members toward patients with mental illness. The critical comments subscale consists of 10 items and is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The critical comments subscale is scored by adding together the ratings from the individual items. Possible scores ranging from 10 to 40 with higher scores indicating greater levels of critical comments with their loved one.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.14 (0.17) |

20. Secondary Outcome: Mean Change in Family Questionnaire of Expressed Emotion - Emotional Overinvolvement (EOI) Subscale
Description: The Family Questionnaire (FQ) is a 20-item, self-administered questionnaire that measures expressed emotion status (criticism and emotional over involvement (EOI)) of family members toward patients with mental illness. The EOI subscale consists of 10 items with each item is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The EOI subscale is scored by adding together the ratings from the individual items. Possible scores ranging from 10 to 40 with higher scores indicating greater levels of emotional overinvolvement with their loved one.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | -0.10 (0.18) |

21. Secondary Outcome: Mean Change in General Health Questionnaire (GHQ) -12 Score - Total Score
Description: The GHQ-12 is a 12-item scale. Answers are on a 4-point scale ranging from 0 "not at all" to 3 "much more than usual." Possible scores range from 0 to 36. Higher scores reflect worse outcomes (more frequent depressive symptoms).
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | -0.48 (0.21) |

22. Secondary Outcome: Mean Change in the Brief Coping Orientation to Problems Experienced (COPE) Scale - Problem-Focused Subscale
Description: The Brief-COPE is a 28-item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. The problem-focused subscale is 8 items. Answers are on a 4-point scale ranging from 1 "I haven't been doing this at all" to 4 "I have been doing this a lot." Possible scores range from 8 to 32. Higher scores on each reflect more frequent use of problem focused coping.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled into the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.46 (0.84) |

23. Secondary Outcome: Mean Change in the Brief Coping Orientation to Problems Experienced (COPE) Scale - Avoidant-Focused Subscale
Description: The Brief-COPE is a 28-item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. The avoidant-focused subscale is 8 items. Answers are on a 4-point scale ranging from 1 "I haven't been doing this at all" to 4 "I have been doing this a lot." Possible scores range from 8 to 32. Higher scores on each reflect more frequent use of avoidance for coping.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled into the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.48 (0.47) |

24. Secondary Outcome: Mean Change in the Brief Coping Orientation to Problems Experienced (COPE) Scale - Emotion-Focused Subscale
Description: The Brief-COPE is a 28-item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. The emotion-focused subscale is 12 items. Answers are on a 4-point scale ranging from 1 "I haven't been doing this at all" to 4 "I have been doing this a lot." Possible scores range from 12 to 48. Higher scores on each reflect more frequent use of emotion focused coping.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled into the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 1.18 (0.81) |

25. Secondary Outcome: Mean Change in Self-Compassion Scale: Short Form (SCS) - Total Score
Description: The Self-Compassion Scale is a 12-item self-report questionnaire designed to measure an individual's self-compassion towards themselves as well as their feelings and emotions. It can be divided into six subscales with two questions for each: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, Over-identified. Answers are on a 5-point scale ranging from 1 "Almost never" to 5 "Almost always." Total score is calculated by totaling the mean of each subscales and reversing the negative subscales (self-judgment, isolation, and over-identification) then taking the mean of the summed subscales. Possible scores range from 1 to 5 with higher scores indicate increased self-compassion.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.33 (0.2) |

26. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Total Score
Description: The Five Facet Mindfulness Questionnaire: 24-item is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. It can be divided into five subscales: Observing, Describing, Acting in Awareness, Non-judging, and Non-reactivity. Answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 24 to 120 once necessary questions (i.e., negative) have been reversed scored. Higher scores indicate more mindfulness and self-awareness.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | -0.47 (1.48) |

27. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Observation Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The observation subscale is 3 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 3 to 15 with higher scores indicate more observational awareness.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | -.039 (0.52) |

28. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Description Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The description subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 after reverse scoring of appropriate items with higher scores indicate more to describe their feelings and experiences.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | -0.50 (0.46) |

29. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Mindful Action Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The mindful action subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 after appropriate items have been reversed scored with higher scores indicate more awareness around their actions and experiences.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | -0.06 (0.46) |

30. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Non-Judgmental Inner Experience Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The non-judgemental subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 once appropriate items have been reversed scored with higher scores indicate more nonjudgmental thoughts towards their beliefs and feelings.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.42 (0.58) |

31. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Non-Reactivity Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The non-reactivity subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 with higher scores indicate more mindful non-reactivity to thoughts and feelings.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | 0.08 (0.57) |

32. Secondary Outcome: Mean Change in the Modified Psychosis Attitude Survey - Total Score
Description: The Modified Psychosis Attitudes Survey is a 19-item self-report questionnaire designed to measure an individual's beliefs and attitude towards psychosis (e.g., identifying psychosis, interacting with individuals experiencing psychosis, etc.). The survey can be divided into 4 subscales: perceived confidence, optimism, fulfillment, and stress-vulnerability orientation. Answers range from "Very strongly disagree", "Strongly disagree", "Mildly disagree", "Neutral", "Mildly agree", "Strongly agree", "Very strongly agree". Total score is obtained with summing each question, after reverse scoring appropriate questions. Possible scores range from 19 to 133. Higher total score indicates an increased knowledge, optimism, and attitudes towards psychosis.
Time Frame: Baseline, Post Treatment (Month 6)
Population: No participants were enrolled in the Treatment as Usual Arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition | Treatment as Usual
Number analyzed (Participants) | 24 | 0
score on a scale | -0.01 (0.17) |

33. Other Pre Specified Outcome: Mean Change in the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure of the 20 DSM-5 symptoms of Post Traumatic Stress Disorder (PTSD). Included in the scale are four domains consistent with the four criteria of PTSD in DSM-5: Re-experiencing (criterion B), Avoidance (criterion C), Negative alterations in cognition and mood (criterion D), and Hyper-arousal (criterion E). Answers are on a 5-point scale including "Not at all," "A little bit," "Moderately," "Quite a bit," and "Extremely" and with total scores ranging from 0 to 80. Higher scores on the PCL-5 reflect more severe trauma-related symptoms.
Time Frame: Baseline, Post Treatment (Month 6)
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Mean Change in the Posttraumatic Growth Inventory (PTGI) Score
Description: The PTGI is a 25-item self-report measure that assesses five domains of personal growth that may follow a stressful encounter. Answers are on a 6-point scale ranging from 0 "I did not experience this" to 5 "I experienced this change to a very great degree." Total scores on this scale range from 0 to 125. Higher scores reflect more positive changes in an individual's life following a stressful experience.
Time Frame: Baseline, Post Treatment (Month 6)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through the post-treatment visit assessment, a total of 6 months.
Description: No participants were enrolled into the Treatment as Usual Arm.
Arm/Group | Altitudes Condition | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/0
Other Adverse Events (participants affected / at risk) | 0/24 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT06094647/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT06094647/ICF_000.pdf